CLINICAL TRIAL: NCT04094064
Title: Evaluation of Accuracy of Continuous Glucose Monitoring (CGM) in Patients With End Stage Renal Disease (ESRD) on Intermittent Hemodialysis (iHD).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Meaghan Stumpf, MD, Assistant Professor, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 190012
Record Dates: First submitted 2019-09-16; First posted 2019-09-18 (Actual); Results first posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-11

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
Keywords: Dialysis; Hemodialysis; Diabetes; Continuous Glucose Monitor (CGM)
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- CGM Use while on Hemodialysis Therapy (Experimental): All subjects will use a CGM for 10 days. Subjects will continue their standard of care hemodialysis treatments during the study period.
  Interventions: Device: Continuous Glucose Monitor

INTERVENTIONS:
Device: Continuous Glucose Monitor — Use of a continuous glucose monitor during study period.

SUMMARY:
Recent advances in continuous glucose monitors (CGMs) and availability of commercial CGM products to patients with type 1 and type 2 diabetes has made the use of CGM more widespread. CGMs work by placing a probe underneath the skin of a patient, into the interstitial space. Patients with end stage renal disease (ESRD) who are on intermittent hemodialysis (iHD) or peritoneal dialysis (PD) undergo fluid shifts between the interstitial fluid and intravascular space during dialysis treatments.These fluid shifts, uremia, acidosis, and volume overload (increase in interstitial fluid volume due to ESRD) have the potential to impact the performance of the most advanced and commercially available CGMs; however, use of CGM in these patients has not yet been studied.Use of CGM, and potentially hybrid closed loop insulin delivery systems that are dependent on accurate continuous glucose monitoring, has the potential to improve glucose control and quality of life in these patients (7). This study team feels that this study will be valuable in collecting preliminary data needed with the goal of validating the use of CGM in this patient population. The specific aim is to conduct a pilot study to evaluate the accuracy of continuous glucose monitors (CGM) in End Stage Renal Disease (ESRD) patients on intermittent hemodialysis (iHD).

DETAILED DESCRIPTION:
Recent advances in continuous glucose monitors (CGMs) and availability of commercial CGM products to patients with type 1 and type 2 diabetes has made the use of CGM more widespread (1). CGMs work by placing a probe underneath the skin of a patient, into the interstitial space. The probe is an electroenzymatic sensor which uses glucose oxidase to break down glucose to create hydrogen peroxidase and other elements. Hydrogen peroxidase then interacts with a base metal layer of the sensor and is oxidized, which results in release of electrons which creates a current. The current is proportional to the glucose concentration. The current is measured by the probe and transmits a calculated glucose concentration to a receiving device (2). Substances that are widely distributed in body water, and thereby present in the interstitial space, potentially affect this technology. Acetaminophen and aspirin are substances that are have been known to affect the accuracy of these devices (3); however, more recently developed CGMs such as the Dexcom G6, were able to demonstrate no interference by acetaminophen (4). Patients with end stage renal disease (ESRD) who are on intermittent hemodialysis (iHD) or peritoneal dialysis (PD) undergo fluid shifts between the interstitial fluid and intravascular space during dialysis treatments. They are also often uremic and have metabolic acidosis (5). These fluid shifts, uremia, acidosis, and volume overload (increase in interstitial fluid volume due to ESRD) have the potential to impact the performance of the most advanced and commercially available CGMs; however, use of CGM in these patients has not yet been studied (3). Moderate to severe CKD is associated with both increase in insulin resistance and decrease in insulin clearance, which results in often unpredictable and labile glucose concentrations and increased risk of hypoglycemia in these patients (6). Use of CGM, and potentially hybrid closed loop insulin delivery systems that are dependent on accurate continuous glucose monitoring, has the potential to improve glucose control and quality of life in these patients (7). This study team feels that this study will be valuable in collecting preliminary data needed with the goal of validating the use of CGM in this patient population.OBJECTIVE: The specific aim is to conduct a pilot study to evaluate the accuracy of continuous glucose monitors (CGM) in End Stage Renal Disease (ESRD) patients on intermittent hemodialysis (iHD). Accuracy will be assessed by calculating the mean absolute relative difference (MARD) between CGM values and concurrent finger stick or capillary blood glucose (CBG) in these patients during hemodialysis, and on non-dialysis days.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18+
* Type 1 diabetes mellitus on intermittent HD thrice weekly OR Type 2 diabetes mellitus on intermittent HD thrice weekly
* Willingness and ability to comply with scheduled visits and study procedures

Exclusion Criteria:

* Inability to comply with finger stick blood glucoses at least four times daily
* Noncompliant with HD therapies
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meaghan Stumpf, MD, Principal Investigator — University of Virginia
Locations (1):
- Meaghan Stumpf, MD, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
There are no current plans to share IPD for this study.

REFERENCES:
- [Result] Villard O, Breton MD, Rao S, Voelmle MK, Fuller MR, Myers HE, McFadden RK, Luke ZS, Wakeman CA, Clancy-Oliveri M, Basu A, Stumpf MM. Accuracy of a Factory-Calibrated Continuous Glucose Monitor in Individuals With Diabetes on Hemodialysis. Diabetes Care. 2022 Jul 7;45(7):1666-1669. doi: 10.2337/dc22-0073. PMID 35485908

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants for this feasibility pilot study were recruited from three University of Virginia Hemodialysis Clinics - Charlottesville, Lynchburg, and Zion's Crossroads between February 2020 through September 2021.
Pre-assignment Details: Participants were approached during their regularly scheduled dialysis session. Upon consent, inclusion/exclusion criteria, medical history and medications were assessed. A serum pregnancy test was performed for women who were of child-bearing potential (negative result required). Eligible participants continued with the continuous glucose monitor (CGM) Pro training visit on the same day or at a later date.
Groups:
- CGM Use While on Hemodialysis Therapy: Participants enrolled in the study wore a blinded Dexcom G6 Pro CGM placed for 10 days which measured the interstitial glucose and recorded interstitial blood glucose every 5 minutes. The participants also checked venous blood glucose values (SMBGs) using a provided study blood glucometer seven times daily on non-hemodialysis (HD) days. During HD sessions, a study team member measured blood glucose with the use of an i-STAT System point of care machine approximately 10-12 times at the following intervals: q15 minutes x 90 minutes, q30 minutes x 60 minutes, then q60 minutes until HD finished. The results from the i-STAT System glucose measurements were recorded in a study flowsheet. The study glucometers recorded and stored the results of SMBG values that were collected each day (10 days) after placement of the sensor.
Period: Overall Study
Arm/Group | CGM Use While on Hemodialysis Therapy
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- CGM Use While on Hemodialysis Therapy: Participants enrolled in the study wore a blinded CGM placed for 10 days which measured the interstitial glucose and recorded interstitial blood glucose every 5 minutes. The participants also checked venous blood glucose values (SMBGs) using a provided study blood glucometer seven times daily on non-hemodialysis (HD) days. During HD sessions, a study team member measured blood glucose with the use of an i-STAT System point of care machine approximately 10-12 times at the following intervals: q15 minutes x 90 minutes, q30 minutes x 60 minutes, then q60 minutes until HD finished. The results from the i-STAT System glucose measurements were recorded in a study flowsheet. The study glucometers recorded and stored the results of SMBG values that were collected each day (10 days) after placement of the sensor.
Arm/Group | CGM Use While on Hemodialysis Therapy
Number analyzed (Participants) | 20
Age, Customized [Mean (Standard Deviation); unit: years] | 60.2 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Diabetes Diagnosis [Count of Participants; unit: Participants]
  Type 1 Diabetes | 4
  Type 2 Diabetes | 15
  Post-Transplantation Diabetes | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Absolute Relative Difference Between CGM Value and Capillary Blood Glucose (Self-monitoring Blood Glucose [SMBG])
Description: Mean Absolute Relative Difference (MARD) between CGM value and capillary blood glucose (SMBG) performed at home 4 to 7 times per day by the participant for 684 matched pairs.
Time Frame: From CGM placement to CGM removal (10 days)
Measure: Mean (Inter-Quartile Range); unit: percent difference
Units Other Than Participants: Overall Matched Pairs
Groups:
- MARD (%): Self-Monitoring Blood Glucose (SMBG): Mean Absolute Relative Difference (MARD) between CGM value and capillary blood glucose (SMBG) performed at home 4 to 7 times per day by the participant for 684 matched pairs.
Arm/Group | MARD (%): Self-Monitoring Blood Glucose (SMBG)
Number analyzed (Participants) | 20
Number analyzed (Overall Matched Pairs) | 684
percent difference | 13.8 [4.9 to 18.2]

2. Primary Outcome: Mean Absolute Relative Difference (MARD) Between Continuous Glucose Monitor (CGM) Value and Venous Blood Glucose (vBGM)
Description: Venous blood glucose samples were collected approximately 12 blood samples from the existing hemodialysis (HD) intravenous (IV) line during each (three) HD session the CGM sensor was worn. These blood samples were immediately processed using the i-STAT System. While the goal was to have the subject participate in three hemodialysis sessions, two sessions were acceptable. 624 matched data pairs were analyzed.
Time Frame: From CGM placement to CGM removal (10 days)
Measure: Mean (Inter-Quartile Range); unit: percent difference
Units Other Than Participants: Overall Matched Pairs
Arm/Group | CGM Use While on Hemodialysis Therapy
Number analyzed (Participants) | 20
Number analyzed (Overall Matched Pairs) | 624
percent difference | 14.3 [5.0 to 19.7]

ADVERSE EVENTS:
Time Frame: Data was recorded once continuous glucose monitor was placed on study participant and until the removal of the continuous glucose monitor (10 days).
Arm/Group | CGM Use While on Hemodialysis Therapy
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-04): https://cdn.clinicaltrials.gov/large-docs/64/NCT04094064/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/64/NCT04094064/ICF_001.pdf